CLINICAL TRIAL: NCT06112015
Title: Effect of Trunk Position on Muscle Activations During Traditional and Suspension Based Bulgarian Split Squat
Brief Title: Muscle Activations During Bulgarian Split Squat Exercise Variations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: Gazi University (Other)
Responsible Party: Principal Investigator, Elif AYGUN POLAT, Principal Investigator, Ordu University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: ODU-SBFTR-AYGUNPOLAT
Record Dates: First submitted 2023-10-19; First posted 2023-11-01 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Sports Physical Therapy
Keywords: Electromyography; Exercise Theraphy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- female athletes (Experimental): 21 female athletes from different branches performed 4 different sessions of Bulgarian split squat exercises.
  Interventions: Other: Bulgarian split squat exercise variations

INTERVENTIONS:
Other: Bulgarian split squat exercise variations — The participants performed 4 different sessions of Bulgarian split squat exercises-Bulgarian split squat with trunk flexion (BSS flexion), Bulgarian Split squat with trunk neutral (BSS neutral), suspension based Bulgarian split squat with trunk flexion (SBSS flexion), suspension based Bulgarian split squat with trunk neutral (SBSS neutral)-with EMG recordings being taken from the dominant extremity throughout each session. For each exercise, participants were instructed to perform three successful repetitions. Between each repetition, there was a 30-second break, and there was at least 10 minutes in between each of the 4 exercises. The movement was standardized by a metronome. The modified Borg scale was used to ensure that fatigue did not occur before each exercise since it was believed that fatigue could affect exercise performance. When scores reported using the modified Borg scale were 1 or lower, exercise recording was started.

SUMMARY:
It is essential to practice and train appropriate activation techniques to ensure optimum strength development. Knowing the effects of exercise variations that will minimize the tension forces acting on the knee by increasing the activation of the lumbo-pelvic-hip complex muscles, which are critical during sports activities, is extremely important in terms of preventing injuries. The aim of this study is to compare muscular activations during traditional and suspension-based Bulgarian split squat exercises and to examine the effect of trunk position on muscular activations.

DETAILED DESCRIPTION:
This study utilized a single-group repeated-measures design, where 4 conditions-Bugarian split squat with trunk flexion (BSS flexion), Bulgarian Split squat with trunk neutral (BSS neutral), suspension based Bulgarian split squat with trunk flexion (SBSS flexion), suspension based Bulgarian split squat with trunk neutral (SBSS neutral)-were examined.Participants had to make two separate trips to the lab in order to be accepted into the study. All exercises were introduced to participants at the initial visit. Prior to beginning the exercises on the second visit, the participants' maximum voluntary isometric contraction (MVIC) values were calculated. The muscle activity of the gluteus medius (GMed), gluteus maximus (GMax), vastus lateralis (VL), rectus femoris (RF), vastus medialis (VM), semitendinosus (ST), biceps femoris (BF),and erector spina (ES) was monitored through the root mean square surface EMG signal amplitude. The order of the tasks was chosen for each person by straightforward randomization (by selecting from a deck of shuffled cards) so order to reduce the impact of the sequence of the exercises.The modified Borg scale was used to ensure that fatigue did not occur before each exercise since it was believed that fatigue could affect exercise performance.

ELIGIBILITY:
Inclusion Criteria:

* Being a licensed athlete in one's own field,
* Having been engaged in sports for at least 2 years

Exclusion Criteria:

* Individuals with any musculoskeletal injury history in the lower extremities and trunk that could impede exercise within the last year,
* Individuals with systemic, neurological, and/or cognitive issues,
* Individuals experiencing pain in the lower extremities and trunk during exercises

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-05-30 (Actual)

PRIMARY OUTCOMES:
Surface EMG Measurement | in an average of one hour
  During data collection, the EMG Noraxon MiniDTS system (Noraxon Inc.) was used to measure the signals from the muscle. Additionally, the participants were video-recorded to prevent any potential mistakes that might have gone unnoticed during the activities.
Normalization of Surface EMG | in an average of one hour
  To normalize the EMG data obtained during the exercises, MVIC was performed for each muscle.
  Participants were asked to warm up on a treadmill at submaximal speed for 8 minutes before starting the measurements. Measurements were performed with 3 repetitions, each lasting 5 seconds, and a 1-minute rest period between repetitions. During the measurements, participants were verbally encouraged to give their maximum effort. After the MVIC measurements, participants were given a 5-minute rest period.

CONTACTS AND LOCATIONS:
Overall Officials: Elif AYGUN POLAT, Principal Investigator — Ordu University; Nevin A. GUZEL, Study Director — Gazi University; Sonay GURUHAN, Principal Investigator — Gazi University; Nihan KAFA, Principal Investigator — Gazi University
Locations (1):
- Ordu University, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Aygun-Polat E, Guzel NA, Guruhan S, Polat Y, Karatas N. Targeted muscle activation in Bulgarian split squat variations: effects of trunk position and suspension-based execution. BMC Sports Sci Med Rehabil. 2025 Aug 27;17(1):251. doi: 10.1186/s13102-025-01306-z. PMID 40867012